CLINICAL TRIAL: NCT02351245
Title: Clinical Characteristics and Complications of Infantile Hemangiomas Located in Lips
Brief Title: Clinical Characteristics of Lip Hemangiomas
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Linlin Li, Department of Dermatology, Zhujiang Hospital of Southern Medical University, Zhujiang Hospital
Other Study IDs: IH201412
Record Dates: First submitted 2015-01-19; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Hemangioma
MeSH Terms: conditions — Hemangioma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lip hemangiomas
  Interventions: Other: observation

INTERVENTIONS:
Other: observation

SUMMARY:
Lip hemangiomas are at higher risk than those located in other sites. However, studies about clinical characteristics of lip hemangiomas have not been enough. The investigators want to conduct a prospective study on the clinical features of lip hemangiomas.

DETAILED DESCRIPTION:
Hemangiomas involving lip are of special concern, since they occur in a prominent location on the face and can distort lip anatomy and lead to disfunction. Infantile hemangiomas in lip had significantly higher incidence than the others. It is often difficult to decide which patient with an lip hemangioma is at higher risk.

The investigators are interested in conducting a study on the clinical features of lip hemangiomas. The investigators are collecting medical records and photos of lip hemangiomas, including demographic information, maternal process, birth, location, size and complication. Based on the data, sum up the main points of clinical characteristics and complication.

ELIGIBILITY:
Inclusion Criteria:

* Only lip hemangiomas visiting between June 1, 2010 and October 1, 2014 were included in this study, which was defined as any infantile hemangioma covering any part of vermilion.

Exclusion Criteria:

* Perioral hemangiomas which did not involve vermilion were excluded.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All the patients of lip hemangiomas after Dr. Zhang in Dermatology Clinic of Zhujiang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
appearance time, location, size, complication of lip hemangiomas | up to 2 months

SECONDARY OUTCOMES:
demographic information | up to 1 month
maternal specific events | up to 1 month